CLINICAL TRIAL: NCT01555736
Title: A Randomised Double-blind Clinical Trial for Evaluation of Efficacy and Safety of Perennial in Comparison to Preseasonal Grass/Rye Pollen Immunotherapy in Patients Suffering From Seasonal Allergic Rhinitis
Brief Title: Comparison of Perennial and Preseasonal Subcutaneous Immunotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Collaborators: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Principal Investigator, Piotr Kuna, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ne0103AV
Record Dates: First submitted 2012-03-06; First posted 2012-03-15 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: allergic rhinitis; perennial immunotherapy; preseasonal immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — allergovit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- preseasonal immunotherapy scheme (Active Comparator)
  Interventions: Drug: grass (80%) and rye (20%) pollens allergoids
- perennial immunotherapy scheme (Active Comparator)
  Interventions: Drug: grass (80%) and rye (20%) pollens allergoids

INTERVENTIONS:
Drug: grass (80%) and rye (20%) pollens allergoids — comparison of two schemes of immunotherapy - preseasonal and perennial immunotherapy.
  Other Names: Allergovit

SUMMARY:
Specific immunotherapy, which involves the administration of allergic extracts to patients with symptoms of allergic disorder, is the leading therapeutical tool of modern allergology. According to the latest studies immunotherapy not only reduces symptoms' severity but also may modify the course of allergic disease by reducing the risk of new sensitisations and development of more advanced stages of the disease.It has been hypothesized basing on clinical observation that perennial immunotherapy is more effective and safer in comparison to preseasonal immunotherapy. The aim of the study was to compare the effect of perennial and preseasonal immunotherapy on rhinoconjunctivitis symptoms and safety of both treatments.

ELIGIBILITY:
Inclusion Criteria:

1. IgE-mediated seasonal allergic rhinitis with symptoms during the grass and rye pollens season (May, June, July);
2. Symptoms of allergic rhinoconjunctivitis requiring medication during the last season
3. Positive skin prick test to grass and rye pollens only with wheal at least as large as histamine control reaction and diameter > 5mm;
4. For female patients effective contraception and negative pregnancy test results were necessary.

Exclusion Criteria:

1. Previous course of immunotherapy with grass and rye pollens extracts or allergens which are unknown during the last 5 years
2. FEV1 < 80% of predicted
3. Uncontrolled bronchial asthma according to GINA
4. Non-allergic rhinoconjunctivitis
5. Severe acute or chronic diseases, severe inflammatory diseases
6. Autoimmune diseases, immunosuppression, neoplastic diseases
7. Severe psychiatric and psychological disorders including alcohol or drug abuse
8. Contraindication for application of adrenaline;
9. Treatment with beta-blockers
10. Pregnancy or lactation period
11. Females patients seeking to become pregnant
12. Low compliance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2003-01; Primary Completion 2006-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
difference between preseasonal and perennial immunotherapy in area under curve of combined symptom medication score during 1st year of immunotherapy | up to 3 months
  combined symptom medication score was calculated as a sum of rhinoconjunctivitis symptoms and use of rescue medications during pollen season
difference between preseasonal and perennial immunotherapy in area under curve of combined symptom medication score during 2nd year of immunotherapy | up to 3 months
  combined symptom medication score was calculated as a sum of rhinoconjunctivitis symptoms and use of rescue medications during pollen season
difference between preseasonal and perennial immunotherapy in area under curve of combined symptom medication score during 3rd year of immunotherapy | up to 3 months
  combined symptom medication score was calculated as a sum of rhinoconjunctivitis symptoms and use of rescue medications during pollen season

SECONDARY OUTCOMES:
frequency of adverse reactions during immunotherapy | up to 3 years of immunotherapy
type of adverse reactions | up to 3 years of immunotherapy
the differences from baseline in mean daily rhinoconjunctivitis symptoms score | up to 3 months/4 years
the differences between study groups in mean daily rhinoconjunctivitis symptoms score | up to 3 months/4 years
the differences from baseline in combined symptom medication score | up to 3 months/4 years
the differences from baseline a in serum level of sIgG4 | the peak of each pollen season (June) during 4 years of study
the differences between study groups in combined symptom medication score | up to 3 months/4 years
the differences between study groups in serum level of sIgG4 | up to 3 months/4 years

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, MD, PhD, Principal Investigator — Department of Internal Diseases, Asthma and allergy, Medical University of Lodz
Locations (1):
- Department of Internal diseases, Asthma and Allergy, Lodz, Poland

REFERENCES:
- [Derived] Tworek D, Bochenska-Marciniak M, Kuprys-Lipinska I, Kupczyk M, Kuna P. Perennial is more effective than preseasonal subcutaneous immunotherapy in the treatment of seasonal allergic rhinoconjunctivitis. Am J Rhinol Allergy. 2013 Jul-Aug;27(4):304-8. doi: 10.2500/ajra.2013.27.3935. Epub 2013 Apr 29. PMID 23636036